CLINICAL TRIAL: NCT05936385
Title: Mobile Integrated Care for Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Health System (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Thao-Ly Phan, Associate Professor of Pediatrics, Nemours Children's Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 416-Project; P20GM144270 (NIH)
Record Dates: First submitted 2023-06-20; First posted 2023-07-07 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Disparities; Stakeholder engagement; Social determinants of health; Healthcare delivery
MeSH Terms: conditions — Obesity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Lifestyle (Experimental): Healthy lifestyle counseling and goal setting every month with a team of experts, mobile app with healthy lifestyle resources and goal tracking tool, access to social services and lifestyle programs in the community, and community health worker outreach every month.
  Interventions: Behavioral: Healthy Lifestyle
- Standard of Care (Active Comparator): Weight checks and lifestyle counseling with primary care provider every other month.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Healthy Lifestyle — Healthy lifestyle counseling and goal setting every month with a team of experts, mobile app with healthy lifestyle resources and goal tracking tool, access to social services and lifestyle programs in the community, and community health worker outreach every month.
  Arms: Healthy Lifestyle
Behavioral: Standard of Care — Weight checks and lifestyle counseling with primary care provider every other month.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to evaluate a new way of providing healthcare to children with an unhealthy weight.

Families who participate will be assigned by chance to one of two groups. One group will see their child's primary care provider to talk about healthy lifestyles for 6 months.

The other group will be in our Healthy Lifestyle program for 6 months. This will include:

* Check-ins with lifestyle specialists and community health workers,
* A mobile app to help support a healthy lifestyle, and
* Access to community programs and activities.

The main questions the study aims to answer are:

* Do children in the Healthy Lifestyle program have better weight outcomes?
* Do more families in the Healthy Lifestyle program stay in the study?
* Does the Healthy Lifestyle program work better for families from certain communities?

ELIGIBILITY:
Caregiver and child dyads will be enrolled

Inclusion Criteria:

* Child 4-12 years of age
* Child is a patient of the Nemours Children's Health primary care clinics in Milford, Seaford, and Millsboro
* Child has a BMI ≥ 95% for age and sex
* Child is from a clinic serving rural neighborhoods (RUCA ≥ 4)

Exclusion Criteria:

* Caregiver not child's legal guardian
* Caregiver not proficient in English or Spanish
* Caregiver does not have a device and reliable internet
* Child has a genetic syndrome or endocrine disorder that predisposes to obesity
* Child is on a medication that impacts weight
* Child is already enrolled in a weight management program

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thao-Ly T Phan, MD, MPH, Principal Investigator — Nemours Children's Health
Locations (3):
- United States (3):
  - Nemours Children's Health, Milford, Milford, Delaware
  - Nemours Children's Health, Millsboro, Millsboro, Delaware
  - Nemours Children's Health, Seaford, Seaford, Delaware

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Lifestyle | Standard of Care
Started | 29 | 30
Completed | 21 | 22
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Lifestyle | Standard of Care | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.1 (2.5) | 8.2 (2.6) | 8.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 21 | 22 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
BMI percentile above the 95th percentile [Mean (Standard Deviation); unit: BMI percentile above the 95th percentile] — American Academy of Pediatrics guidelines recommend using percentiles of the 95th percentile of BMI-for-age to indicate different levels of severe obesity. More information on the methodology for this can be found at https://www.cdc.gov/growthcharts/extended-bmi-data-files.htm.
  BMI percentile above the 95th percentile | 119.4 (14.2) | 123.9 (19.8) | 121.8 (17.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Adiposity
Description: Change in BMI percentile (above the 95th percentile) for age and sex. Height and weight measurements will be used to calculate BMI percentile above the 95th percentile based on CDC algorithms.
Time Frame: 6 months
Population: 7 participants did not have anthropometric measurements collected in the EHR at the end of study
Measure: Mean (Standard Deviation); unit: Change in BMI percentile
Arm/Group | Healthy Lifestyle | Standard of Care
Number analyzed (Participants) | 25 | 27
Change in BMI percentile | -0.55 (7.18) | 0.64 (5.30)

2. Primary Outcome: Visit Adherence
Description: Lost to follow-up (attrition) from study as documented in the electronic health record.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Lifestyle | Standard of Care
Number analyzed (Participants) | 29 | 30
Participants | 8 | 8

3. Secondary Outcome: Differences in Change in Child Adiposity Based on Child Sociodemographic Characteristics
Description: Differences in change in BMI percentile (above the 95th percentile) for age and sex between subgroups based on race, ethnicity, and insurance status. Height and weight measurements will be used to calculate BMI percentile above the 95th percentile based on CDC algorithms. Child race, ethnicity, and insurance status will be collected from parents at the time of enrollment.
Time Frame: 6 months
Population: 7 participants did not have anthropometric measures recorded in the EHR at baseline and study end due to lost to follow-up
Measure: Mean (Standard Deviation); unit: Change in BMI percentile
Arm/Group | Healthy Lifestyle | Standard of Care
Number analyzed (Participants) | 25 | 27
Change in BMI percentile
  Non-Hispanic White: number analyzed (Participants) | 9 | 10
  Non-Hispanic White | -0.56 (7.11) | -0.09 (6.83)
  Non-Hispanic Black: number analyzed (Participants) | 8 | 11
  Non-Hispanic Black | 0.81 (4.61) | 1.67 (4.38)
  Hispanic or Latino: number analyzed (Participants) | 8 | 6
  Hispanic or Latino | -1.90 (9.68) | -0.04 (4.43)
  Private Insurance: number analyzed (Participants) | 5 | 8
  Private Insurance | -1.64 (2.16) | 0.04 (6.24)
  Public Insurance: number analyzed (Participants) | 20 | 19
  Public Insurance | -0.28 (7.99) | 0.89 (5.02)

4. Secondary Outcome: Differences in Visit Adherence Based on Child Sociodemographic Characteristics
Description: Differences in lost to follow-up (attrition) from study as documented in the electronic health record between subgroups based on race, ethnicity, and insurance status. Child race, ethnicity, and insurance status will be collected from parents at the time of enrollment.
Time Frame: 6 months
Population: Number analyzed in rows below are only those who were lost to follow-up (attrition) for each race, ethnicity, or insurance category
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Lifestyle | Standard of Care
Number analyzed (Participants) | 29 | 30
Participants
  Non-Hispanic Black: number analyzed (Participants) | 10 | 11
  Non-Hispanic Black: Attrition | 5 | 4
  Non-Hispanic Black: Non-Attrition | 5 | 7
  Non-Hispanic White: number analyzed (Participants) | 11 | 11
  Non-Hispanic White: Attrition | 3 | 1
  Non-Hispanic White: Non-Attrition | 8 | 10
  Hispanic or Latino: number analyzed (Participants) | 8 | 8
  Hispanic or Latino: Attrition | 0 | 3
  Hispanic or Latino: Non-Attrition | 8 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Healthy Lifestyle | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT05936385/Prot_SAP_000.pdf